CLINICAL TRIAL: NCT00093678
Title: A Randomized, Double Blind, Placebo-Controlled Trial of Celecoxib in Patients With Advanced Cancer
Brief Title: Celecoxib in Managing Pain, Weight Loss, and Weakness in Patients With Advanced Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000389434; ECOG-E1Z02
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Cachexia; Lymphoma; Melanoma (Skin); Ovarian Cancer; Pain; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: pain; cachexia; unspecified adult solid tumor, protocol specific; recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; ovarian sarcoma; recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent melanoma; stage III melanoma; stage IV melanoma; chondrosarcoma; metastatic osteosarcoma; recurrent osteosarcoma; classic Kaposi sarcoma; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; intraocular lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; primary central nervous system lymphoma; recurrent adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; recurrent mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; immunosuppressive treatment related Kaposi sarcoma
MeSH Terms: conditions — Cachexia; Lymphoma; Melanoma; Ovarian Neoplasms; Pain; Sarcoma; Chondrosarcoma; Osteosarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Waldenstrom Macroglobulinemia; Mycosis Fungoides; Sezary Syndrome; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Celecoxib; Nutritional Support; Analgesia; Palliative Care

INTERVENTIONS:
Drug: celecoxib
Procedure: anticachectic therapy
Procedure: nutritional support
Procedure: pain therapy
Procedure: supportive care/therapy

SUMMARY:
RATIONALE: Celecoxib may help relieve moderate or severe pain associated with cancer. It may also decrease weight loss and improve muscle strength in cancer patients.

PURPOSE: This randomized clinical trial is studying celecoxib to see how well it works in managing pain, weight loss, and weakness in patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the symptom burden and functional status, as measured by the physical well-being subscale of the Functional Assessment of Cancer Therapy-General (FACT-G), of patients with advanced cancer treated with celecoxib vs placebo.

Secondary

* Compare pain, as measured by the Brief Pain Inventory, in patients treated with these drugs.
* Compare the need for opioid analgesics, as measured by the oral morphine equivalent of analgesics used, in patients treated with these drugs.
* Compare weight loss in patients treated with these drugs.
* Compare quality of life, as measured by the FACT-G, in patients treated with these drugs.
* Compare the median survival of patients treated with these drugs.
* Determine the toxicity of celecoxib in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to ECOG performance status (0 or 1 vs 2 or 3), need for opioid analgesics within the past 2 weeks (yes vs no), and weight loss as percentage of baseline body weight (< 5% vs ≥ 5%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral celecoxib twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms, treatment continues in the absence of unacceptable toxicity.

Quality of life is assessed at baseline and at 2, 6, and 12 weeks.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 296 patients (148 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant tumor of 1 of the following types:

  * Carcinoma
  * Sarcoma
  * Melanoma
  * Lymphoma
* Metastatic or unresectable disease
* Clear evidence of residual disease after most recent prior treatment

  * Measurable disease not required
* Patient has elected to receive supportive care only rather than active cancer treatment (e.g., palliative chemotherapy)
* Brain metastases allowed provided the following criteria are met:

  * Completed treatment for CNS disease (e.g., whole brain radiotherapy, surgery, or stereotactic surgery)
  * Clinically stable disease for at least 4 weeks after treatment completion
  * No requirement for corticosteroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* ALT and AST ≤ 5 times ULN

Renal

* Creatinine ≤ 1.6 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No transient ischemic attack within the past 6 months
* No stroke within the past 6 months
* No angina pectoris requiring medical therapy
* No other active coronary artery disease or cerebrovascular disease

Other

* No active gastrointestinal (GI) ulcer disease
* No GI bleeding
* No history of allergic reaction, urticaria, or bronchospasm after taking NSAIDs, aspirin, or sulfonamide drugs
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent hematopoietic growth factors for cytopenia or fatigue allowed
* No concurrent biologic anticancer agents

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics
* No concurrent corticosteroids for management of cancer-related symptoms or other illness
* No concurrent hormonal therapy

  * Concurrent luteinizing hormone-releasing hormone therapy allowed for prostate cancer patients provided drug was initiated at least 6 months ago AND there is unequivocal evidence of progressive disease, defined by 1 of the following criteria:

    * Rising prostate-specific antigen (PSA) on 3 successive measurements
    * Rising PSA on 2 measurements taken at least 2 weeks apart
    * New lesions on bone scan

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Other

* Concurrent bisphosphonates for management of osseous metastases or hypercalcemia allowed
* No concurrent cytotoxic drugs
* No other concurrent nonsteroidal anti-inflammatory drugs (NSAIDs) or aspirin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald P. Lawrence, MD, Study Chair — Tufts Medical Center; Michael J. Fisch, MD, MPH, FACP — M.D. Anderson Cancer Center